CLINICAL TRIAL: NCT04146935
Title: Examining the Effect of Burosumab on Muscle Function Using MR Spectroscopy
Brief Title: Examining the Effect of Burosumab on Muscle Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2000026400
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: X-linked Hypophosphatemia
Keywords: Crysvita; Burosumab
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with XLH (Experimental): Patients will receive Burosumab monthly at visits 1,2 and 3 subcutaneously at a dose of 1.0 mg/kg. Dose may be adjusted as needed.
  Interventions: Drug: Burosumab Injection [Crysvita]

INTERVENTIONS:
Drug: Burosumab Injection [Crysvita] — Burosumab/Crysvita SC injection monthly
  Other Names: Crysvita

SUMMARY:
Patients with X-linked hypophosphatemia (XLH) often report symptoms of fatigue and weakness particularly after exertion, in addition to their skeletal complaints. In previous trials using KRN23 (same drug as burosumab/Crysvita®), patients report these symptoms improve. The investigators wish to test this hypothesis directly by measuring muscle energy when patients begin treatment with Crysvita® for the first time.

DETAILED DESCRIPTION:
X-linked hypophosphatemia is a skeletal dysplasia. The mineralized tissue complications of XLH have been the focus of investigative studies seeking to understand its pathogenesis, as well as studies directed at new therapies. However, in addition to their skeletal complaints, patients with XLH have among their most frequent symptoms, fatigue and weakness, which manifest as both a generalized sense of a lack of energy as well as a more specific feeling that their muscular function is impaired. Objectively, patients complain of fatigue after exertion, when otherwise they do not think they should expect to feel so spent. These symptoms occur in individuals who otherwise have good cardiovascular and respiratory health, so co-morbidities are unlikely to explain these pervasive complaints. Anecdotally, the investigators open-label trial data using KRN23 suggest that these symptoms are dramatically ameliorated by treatment with the drug. In a recent study¹, the investigators found that when stressed by a low-phosphate diet, rates of insulin-stimulated myocyte Adenosine triphosphate (ATP) flux were reduced by 50% in an experimental model of systemic hypophosphatemia (the NaPi2a knockout mouse). Moreover, ATP synthetic flux correlated directly with cellular and mitochondrial phosphate uptake in two rodent myocyte cell lines, as well as in freshly isolated myocyte mitochondria. As direct evidence that these preclinical findings are relevant to human hypophosphatemic genetic syndromes we studied a patient with Heredity Hypophosphatemic Rickets with Hypercalciuria (HHRH) who was not being treated at the time of our experiment. In this patient who had a 50% reduction in serum phosphate, muscle ATP content was also significantly reduced ¹. Both of these parameters normalized completely with oral phosphate repletion ¹. These data strongly support the hypothesis that reduced muscle ATP flux may underlie the myopathy seen in patients with XLH. The investigators propose to directly test this hypothesis, in patients about to begin treatment with Crysvita® for the first time.

Muscle tissue phosphorus concentration and ATP flux rates will be assessed in the right gastrocnemius of the lower leg using 31P-NMR (nuclear magnetic resonance) spectroscopy over the course of the 3 month study. The study consists of 5 visits total over 3 months. At visits 1,4 and 5, patients will undergo magnetic resonance (MR) spectroscopy assessments and functional testing along with blood and urine analysis. At visits 1,2 and 3 patients will receive Burosumab/Crysvita® by subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age
2. Diagnosis of XLH
3. eGFR ≥ 50 (estimated glomerular filtration rate)
4. Normal serum calcium
5. Phosphate ≤ 2.5 mg/dl
6. Deemed clinically appropriate for starting therapy with Burosumab/Crysvita® (based on the treating physician's evaluation)
7. Deemed appropriate for MR Spectroscopy

Exclusion Criteria:

1. Patients with fixed skeletal abnormalities which would prevent them from successfully completing study-related functional assessments
2. Patients unwilling to stop therapy with supplemental phosphate and calcitriol 2 weeks prior to enrollment.
3. Patients who have undergone an orthopaedic procedure within the previous 6 months involving implantation of metal hardware

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl L Insogna, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pesta DH, Tsirigotis DN, Befroy DE, Caballero D, Jurczak MJ, Rahimi Y, Cline GW, Dufour S, Birkenfeld AL, Rothman DL, Carpenter TO, Insogna K, Petersen KF, Bergwitz C, Shulman GI. Hypophosphatemia promotes lower rates of muscle ATP synthesis. FASEB J. 2016 Oct;30(10):3378-3387. doi: 10.1096/fj.201600473R. Epub 2016 Jun 23. PMID 27338702

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With XLH
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With XLH
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
  Canada | 2
Fasting serum phosphate [Mean (Standard Deviation); unit: mg/dL] | 1.74 (0.43)
Serum calcium [Mean (Standard Deviation); unit: mg/dL] | 9.30 (0.32)
Parathyroid hormone (PTH) [Mean (Standard Deviation); unit: pg/mL] | 68.78 (24.40)
Renal phosphate threshold [Mean (Standard Deviation); unit: mg/100 ml GF] | 1.59 (0.44)
Fibroblast growth factor (FGF) 23 levels [Mean (Standard Deviation); unit: pg/mL] | 53.4 (14.5)
25-hydroxy vitamin D [Mean (Standard Deviation); unit: ng/mL] | 34.23 (15.53)
1,25-dihydroxy vitamin D [Mean (Standard Deviation); unit: pg/mL] | 71.29 (19.05)
Serum creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.63 (0.15)

OUTCOME MEASURES:

1. Primary Outcome: Skeletal Muscle Adenosine Triphosphate (ATP) Synthesis Rate
Description: Rates of mitochondrial phosphorylation activity were assessed in the soleus/gastrocnemius muscle complex of the right calf by 31P magnetic resonance spectroscopy saturation transfer technique (micro-mol/g/min)
Time Frame: 2.5 months
Measure: Least Squares Mean (95% Confidence Interval); unit: umol/g/min
Arm/Group | Patients With XLH
Number analyzed (Participants) | 10
umol/g/min | 9.41 [8.7827 to 10.0333]
Statistical Analysis 1: Comparison: Patients With XLH; Test type: Other — Mixed model repeated measures; p = 0.4147, Mixed Models Analysis — Visit 1 (baseline) to visit 4 (peak)

2. Secondary Outcome: Serum Phosphate
Description: measured in mg/dl
Time Frame: 2.5 months
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Patients With XLH
Number analyzed (Participants) | 10
mg/dL | 2.85 [2.4231 to 3.2769]
Statistical Analysis 1: Comparison: Patients With XLH; Test type: Other; p < .0001, Mixed Models Analysis

3. Secondary Outcome: Intracellular Phosphate Concentration in Umol/g Muscle
Description: Intracellular phosphorus concentration in skeletal muscle (umol/g muscle)
Time Frame: 2.5 months
Measure: Least Squares Mean (95% Confidence Interval); unit: umol/g muscle
Arm/Group | Patients With XLH
Number analyzed (Participants) | 10
umol/g muscle | 2.31 [1.9654 to 2.6446]
Statistical Analysis 1: Comparison: Patients With XLH; Test type: Other — Mixed model repeated measures; p = 0.6957, Mixed Models Analysis

4. Other Pre Specified Outcome: Six-minute Walk Test
Description: functional testing outcome measured in meters
Time Frame: 2.5 months
Measure: Least Squares Mean (95% Confidence Interval); unit: meter
Arm/Group | Patients With XLH
Number analyzed (Participants) | 10
meter | 440.4 [388.06 to 492.74]
Statistical Analysis 1: Comparison: Patients With XLH; Test type: Other; p = 0.0092, Mixed Models Analysis

5. Other Pre Specified Outcome: Sit to Stand
Description: functional testing outcome measured in the number completed in 30 seconds
Time Frame: 2.5 months
Measure: Least Squares Mean (95% Confidence Interval); unit: repetitions
Arm/Group | Patients With XLH
Number analyzed (Participants) | 10
repetitions | 14.2 [10.8312 to 17.5688]
Statistical Analysis 1: Comparison: Patients With XLH; Test type: Other — Mixed model repeated measures; p = 0.1383, Mixed Models Analysis

6. Other Pre Specified Outcome: Timed up and go Test
Description: functional testing outcome measured in seconds
Time Frame: 2.5 months
Measure: Least Squares Mean (95% Confidence Interval); unit: second
Arm/Group | Patients With XLH
Number analyzed (Participants) | 10
second | 7.47 [6.4473 to 8.4967]
Statistical Analysis 1: Comparison: Patients With XLH; Test type: Other — mixed model repeated measures; p = 0.0572, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 3 months (time of consent to completion of visit 5)
Arm/Group | Patients With XLH
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With XLH (N=10)
Partial ureteropelvic junction obstruction by staghorn calculus (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT04146935/Prot_SAP_000.pdf